CLINICAL TRIAL: NCT02422680
Title: Patient Satisfaction With Colonoscopy in a Danish Setting - What Are the Most Important Factors?
Status: Withdrawn | Type: Observational
Why Stopped: Cancelled according to PhD-protocol with insufficient time to complete the study
Sponsor: Aalborg University Hospital (Other)
Collaborators: Nordsim (Unknown)
Responsible Party: Principal Investigator, Lasse Pedersen, MD, Ph.D.-student, Aalborg University Hospital
Other Study IDs: AalborgH
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Cancer
Keywords: Quality assurance; Caecum intubation rate; Patient satisfaction
MeSH Terms: conditions — Colorectal Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients referred to a colonoscopy: A min. of 800 patients referred to colonoscopy at Aalborg University Hospital. The 800 patients are from the out patient clinic. A mix of screening and non-screening patients.
  Interventions: Procedure: No intervention, purely observational.

INTERVENTIONS:
Procedure: No intervention, purely observational. — No intervention is made other than following existing guidelines for colonoscopy. Further treatment and/or renewed colonoscopy in case of positive findings follows existing guidelines. The group is used only used to collect quality assurance data.

SUMMARY:
The study aim is to investigate factors associated with patient satisfaction during a colonoscopy.

DETAILED DESCRIPTION:
The study aim to capture key quality indicators and patient satisfaction for 800 patients referred for a colonoscopy at Aalborg University Hospital. The patient population is mix of screening and non-screening colonoscopies seen at our out-patient clinic.

Each Colonoscopy is registered using a specially designed registration form and a more detailed form relating to the colonoscopy itself. The data collected includes: The Colonoscopist endoscopy experience and education, Medicine use, Colonoscopy duration, Unadjusted Caecum Intubations rate, Polyp detection rate, Polyps removed, Cancer detection rate and Nurse assisted Gloucester Comfort score.

Patient level data were recorded using a questionaire with 6 questions regarding satisfaction, pain, discomfort etc on a 10 cm analog scale.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to colonoscopy at the out-patient clinic at Aalborg University department.

Exclusion Criteria:

* Rejection to fill out questionaire.
* Patents referred to AVA (advanced endoscopy unit) were excluded as the are not comparable to regular colonoscopies. Most patients are referred to AVA for specific endoscopy treatments such as large polyp removals etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to colonoscopy at the out patient clinic at Aalborg University department. All patients deemed fit to for at colonoscopy at the outpaient clinic were included. The patient population is a mix of screening and non-screening patients. The study begins in april 2015.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | 1 day
  Each patient were given a questionaire with 6 questions answering satisfaction, pain, discomfort etc on a 10 cm analog scale.

SECONDARY OUTCOMES:
Nurses perception of patients' pain | 1 day
  Nurse assisted Gloucester Comfort score
Patient Pain (own Perception) | 1 day
  10 cm analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Pedersen, m.d., Principal Investigator — Aalborg University Hospital, Surgical Department.
Locations (1):
- NordSim, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chartier L, Arthurs E, Sewitch MJ. Patient satisfaction with colonoscopy: a literature review and pilot study. Can J Gastroenterol. 2009 Mar;23(3):203-9. doi: 10.1155/2009/903545. PMID 19319384